CLINICAL TRIAL: NCT03445117
Title: Increasing the Uptake of Influenza and Pneumococcal Vaccines Among High-Risk Adult Patients Through General Practitioner Clinics
Brief Title: Increasing the Uptake of Influenza and Pneumococcal Vaccines Among High-Risk Adult Patients Through GP Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Frontier Healthcare Group (Unknown); OneCare Medical Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: DSRB 2017/00441
Record Dates: First submitted 2018-01-28; First posted 2018-02-26 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Immunization Programs
Keywords: Influenza Vaccines; Pneumococcal Vaccines; Primary Health Care; Health Communication; Cross-Over Studies; Randomized Controlled Trial
MeSH Terms: conditions — Influenza, Human | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: two-arm cluster randomised crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Clinics assigned to the intervention arm will receive an educational intervention. This comprises posters on vaccination to be put up in the clinic, as well as a flyer which will be handed out by the clinic assistants to all patients 65 years and above, at the point of registration. The poster and flyer content will provide simple messaging to encourage patients to receive influenza and pneumococcal vaccinations and inform them of available healthcare subsidies.
  Interventions: Other: Educational intervention
- Control (No Intervention): Clinics assigned to control arm will run as per their normal operations and not have the interventions implemented.

INTERVENTIONS:
Other: Educational intervention — a) The educational intervention comprises putting up posters on vaccination in the clinic, as well as provision of a specially designed flyer to the clinic, which will be handed out by the clinic assistants to all patients 65 years and above, at the point of registration. The poster and flyer content will provide simple messaging to encourage patients to receive influenza and pneumococcal vaccinations and inform them of available healthcare subsidies. b) Reminders to physicians: The flyers will also serve as physical prompts to physicians to encourage vaccination for their patients. Doctors and clinic staff will also be updated on the study protocol and the recommended adult vaccination schedule before commencement of the study.
  Arms: Intervention

SUMMARY:
Pneumonia and influenza are among the top causes of hospitalisation and death in the elderly. While vaccinations are recommended against these diseases, a large proportion of elderly in the community remain unvaccinated, with approximately only 10% vaccinated for either disease. In this study, the investigators aim to implement an intervention package within GP clinics to increase influenza and pneumococcal vaccination rates, especially among elderly patients with chronic diseases.

DETAILED DESCRIPTION:
Influenza and pneumococcal disease contribute considerably to hospitalisation and mortality in the elderly. While recommended vaccines can reduce disease burden, vaccine uptake remains very low in Singapore, with approximately only 10% of elderly appropriately vaccinated for either disease. Improving vaccine uptake rates could be effected through private sector primary care clinics, which are highly accessible in Singapore. An intervention bundle we piloted in one clinic comprised physician reminders and patient-targeted posters and brochures. Influenza and pneumococcal vaccine rates both increased by >30% over the baseline, although half of eligible patients remained unvaccinated. There is thus scope to devise a more effective intervention bundle and demonstrate its efficacy through a more robust and generalisable study design.

This study aims to evaluate the efficacy of an intervention bundle deployed in general practice clinics to promote influenza and pneumococcal vaccine uptake among elderly patients. The intervention bundle components include educational materials such as posters and flyers, which also serve as reminder slips for attending physicians. The intervention will be implemented in a two-arm cluster randomised crossover trial in up to 30 primary care clinics. Control arm clinics will receive no interventions. Clinics will be randomised into either of the two arms for a period of 3 months, followed by a washout of 1 month before a crossover is performed. The investigators will subsequently compare vaccination rates during intervention and control periods to provide evidence for effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen at GP clinics involved in our study AND
* Aged 65 years and above, with or without chronic disease

Exclusion Criteria:

* Patients not seen at GP clinics involved in our study
* Patients aged below 65 years old

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8837 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Difference in influenza vaccination uptake rate for clinics between intervention and non-intervention periods | 8 months (post-study completion)
  The proportion of all eligible patients arriving at each clinic who receive influenza vaccine during the intervention period compared to the non-intervention period for each clinic.
Difference in pneumococcal vaccination uptake rate for clinics between intervention and non-intervention periods | 8 months (post-study completion)
  The proportion of all eligible patients arriving at each clinic who receive pneumococcal vaccine during the intervention period compared to the non-intervention period for each clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Hanley Ho, Principal Investigator — Tan Tock Seng Hospital
Locations (2):
- Singapore (2):
  - Frontier Healthcare Group, Singapore
  - OneCare Medical Group, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho HJ, Tan YR, Cook AR, Koh G, Tham TY, Anwar E, Hui Chiang GS, Lwin MO, Chen MI. Increasing Influenza and Pneumococcal Vaccination Uptake in Seniors Using Point-of-Care Informational Interventions in Primary Care in Singapore: A Pragmatic, Cluster-Randomized Crossover Trial. Am J Public Health. 2019 Dec;109(12):1776-1783. doi: 10.2105/AJPH.2019.305328. Epub 2019 Oct 17. PMID 31622142